CLINICAL TRIAL: NCT01295632
Title: Phase I Parallel Protocol of MK-8669 (Ridaforolimus) + MK-2206 and MK-8669 (Ridaforolimus) + MK-0752 Doublets (MK-MK) in Patients With Advanced Cancer
Brief Title: Safety and Tolerability of Different Dose Combinations of Ridaforolimus With MK-2206 or MK-0752 for Participants With Advanced Cancer (MK-8669-049)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 8669-049
Record Dates: First submitted 2011-02-09; First posted 2011-02-14 (Estimated); Last update posted 2015-08-27 (Estimated); Status verified 2015-08

CONDITIONS: Advanced Cancer
Keywords: Recurrent glioblastoma multiforme; Hormone resistant prostate cancer; Relapsed ovarian carcinoma; Refractory ovarian carcinoma; Refractory breast cancer; Relapsed breast cancer
MeSH Terms: conditions — Glioblastoma; Ovarian Neoplasms; Breast Neoplasms | interventions — ridaforolimus; 3-(4-((4-chlorophenyl)sulfonyl)-4-(2,5-difluorophenyl)cyclohexyl)propanoic acid; MK 2206

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (10):
- Ridaforolimus 20 mg + MK-2206 90 mg (Experimental)
  Interventions: Drug: ridaforolimus; Drug: MK-2206
- Ridaforolimus 20 mg + MK-2206 135 mg (Experimental)
  Interventions: Drug: ridaforolimus; Drug: MK-2206
- Ridaforolimus 30 mg + MK-2206 90 mg (Experimental)
  Interventions: Drug: ridaforolimus; Drug: MK-2206
- Ridaforolimus 30 mg + MK-2206 135 mg (Experimental)
  Interventions: Drug: ridaforolimus; Drug: MK-2206
- Ridaforolimus 30 mg + MK-2206 200 mg (Experimental)
  Interventions: Drug: ridaforolimus; Drug: MK-2206
- Ridaforolimus 40 mg + MK-2206 135 mg (Experimental)
  Interventions: Drug: ridaforolimus; Drug: MK-2206
- Ridaforolimus 40 mg + MK-2206 200 mg (Experimental)
  Interventions: Drug: ridaforolimus; Drug: MK-2206
- Ridaforolimus 20 mg + MK-0752 1800 mg (Experimental): No longer recruiting as of 19 July 2012
  Interventions: Drug: ridaforolimus; Drug: MK-0752
- Ridaforolimus 30 mg + MK-0752 1800 mg (Experimental): No longer recruiting as of 19 July 2012
  Interventions: Drug: ridaforolimus; Drug: MK-0752
- Ridaforolimus 40 mg + MK-0752 1800 mg (Experimental): No longer recruiting as of 19 July 2012
  Interventions: Drug: ridaforolimus; Drug: MK-0752

INTERVENTIONS:
Drug: ridaforolimus — 10 mg enteric-coated tablets, orally, starting dose 2 tablets and escalating to 4 tablets each day for 5 days per week.
  Other Names: MK-8669
Drug: MK-0752 — 300 mg capsule, orally, 6 capsules per dose, once each week.
  Arms: Ridaforolimus 20 mg + MK-0752 1800 mg; Ridaforolimus 30 mg + MK-0752 1800 mg; Ridaforolimus 40 mg + MK-0752 1800 mg
Drug: MK-2206 — Tablets (5 mg, 25 mg, and 200 mg) to equal starting dose of 90 mg and escalating to 200 mg per dose, orally, once each week.
  Arms: Ridaforolimus 20 mg + MK-2206 135 mg; Ridaforolimus 20 mg + MK-2206 90 mg; Ridaforolimus 30 mg + MK-2206 135 mg; Ridaforolimus 30 mg + MK-2206 200 mg; Ridaforolimus 30 mg + MK-2206 90 mg; Ridaforolimus 40 mg + MK-2206 135 mg; Ridaforolimus 40 mg + MK-2206 200 mg

SUMMARY:
This is a two part study of the drug MK-8669 (ridaforolimus) given with MK-2206 or MK-0752. In Part A of the study, the preliminary maximum tolerated dose (MTD) of the drug combinations will be found by giving sequentially higher doses of the study drugs. An expansion cohort of participants may be enrolled to confirm the MTD. New cohorts at other dose levels may be enrolled, depending on the rate of dose limiting toxicities (DLTs) in the planned cohorts. In Part B, an assessment of the efficacy of the drug combinations against selected advanced cancers will be made so that a recommended dose to be used in Phase 2 studies (RPTD) can be found. As of 19 July 2012 the MK-0752 arms of the study were fully enrolled and closed to further recruitment. As of 30 November 2012, no additional participants with prostate cancer will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

Part A of the Study:

Participant must have a histologically-confirmed metastatic or locally advanced solid tumor that has failed to respond to standard therapy, progressed despite standard therapy, or for which standard therapy does not exist. Non Hodgkin Lymphoma (NHL) participants (in Part A only), must have histologically confirmed relapsed/refractory NHL. There is no limit on the number of prior treatment regimens.

Part B of the Study:

* Participant must have performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) Performance Scale.
* Participant must have adequate organ function.
* Participants must be willing to use effective methods of contraception.
* Participant is able to swallow capsules and has no surgical or anatomical condition that will preclude the participant from swallowing and absorbing oral medications on an ongoing basis.
* Participant has no history of a prior malignancy with the exception of cervical intraepithelial neoplasia; basal cell carcinoma of the skin; adequately treated localized prostate carcinoma with Prostate-Specific Antigen (PSA) <1.0; or who has undergone potentially curative therapy with no evidence of that disease for five years, or who is deemed at low risk for recurrence by his/her treating physician.
* Participant has at least one measurable recurrent or metastatic lesion (if a solitary lesion, histological/cytological confirmation of its neoplastic nature is required) with the exception of prostate cancer participants which do not require measurable disease if participant has PSA level of >10 ng/mL.
* Participant must agree to provide archival or newly-obtained tumor tissue sample.

  * Ridaforolimus + MK-2206 Treatment Arm:

    * Participant must have a histologically-confirmed prostate cancer that is refractory to hormone therapy and for which the participant received any number of prior treatment regimens (no longer recruiting as of 30 November 2012), OR
    * Participant must have a histologically-confirmed breast cancer for which the participant received any number of prior treatment regimens. Archival or fresh tissue must demonstrate a low RAS-gene signature and a high Ki67 index label if estrogen receptor (ER)+
  * Ridaforolimus + MK-0752 Treatment Arm:

    * Participant must have a histologically-confirmed recurrent (either primary or secondary) glioblastoma multiforme with radiographic evidence of progression/recurrence of disease, and up to 2 prior treatment regimens for their recurrent disease, and no prior treatment with bevacizumab, OR
    * Participants must have a histologically-confirmed relapsed or refractory ovarian cancer for which the participant received no more than 2 prior treatment regiments which was either relapsed or refractory to the first line treatment.

Exclusion Criteria:

* Participant has had chemotherapy or radiotherapy within 4 weeks prior to study Day 1 (6 weeks for nitrosoureas, mitomycin C), biological therapy (excluding antibodies) within 2 weeks prior to study Day 1, or who has not recovered (≤Grade 1 or baseline) from adverse events due to agents administered more than 4 weeks earlier. Luteinizing-hormone releasing hormone (LHRH) use by prostate cancer patients is permitted; participants with prostate cancer previously treated with flutamide or nilutamide require 4 week washout period and participants previously treated with bicalutamide require 6 week washout period before study drug administration.
* Participant is currently participating or has participated in a study with an investigational compound or device within 28 days, or 5X half-life of the investigational compound (not including monoclonal antibodies), whichever is longer, of Day 1 of this study.
* Participants with known symptomatic or progressing Central Nervous System (CNS) metastases and/or carcinomatous meningitis are excluded. However, participants with CNS metastases who are asymptomatic and have completed a course of therapy are eligible for the study provided they are clinically stable for 1 month prior to entry as defined as: (1) no evidence of new or enlarging CNS metastasis (2) off steroids or on a stable dose of steroids.
* Participant has known hypersensitivity to the components of study drug or its analogs.
* Participant has prior exposure to agents that have the same target as to the study drug.
* Participant has significant or uncontrolled cardiovascular disease, including New York Heart Association (NYHA) Class III-IV heart failure, unstable angina, or a myocardial infarction within the last 6 months.
* Participant is a known diabetic participant who is poorly controlled at screening.
* Participant has known psychiatric or substance abuse disorders that would interfere with compliance with study requirements.
* Participant is, at the time of signing informed consent, a regular user (including "recreational use") of any illicit drugs or had a recent history (within the last year) of drug or alcohol abuse.
* Participant is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the study.
* Participant is known to be Human Immunodeficiency Virus (HIV)-positive.
* Participant has active Hepatitis B or C.
* Participant has symptomatic ascites or pleural effusion. A participant who is clinically stable following treatment for these conditions is eligible.
* Participant has a requirement for concurrent treatment with immunosuppressive agents other than prescribed corticosteroids at stable doses for ≥ 2 weeks prior to first planned dose of study drug.
* Participant has a requirement for concurrent treatment with medication(s) that strongly or moderate induce or inhibit cytochrome P450 (CYP3A). Participants should be off these medications ≥ 2 weeks prior to the first dose of study medication.

  * For participants with glioblastoma, dexamethasone should be discontinued at least 1 week prior to the first dose of study drugs.

For participants on the Ridaforolimus + MK-0752 treatment arm:

- Participant requires or anticipated to require concomitant therapy with enzyme-inducing antiepileptic therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2011-02; Primary Completion 2013-12 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Number of participants receiving ridaforolimus + MK-2206 who experience dose-limiting toxicities (DLTs). | Cycle 1 (28 days)
Number of participants receiving ridaforolimus + MK-0752 who experience DLTs. | Cycle 1 (28 days)
Number of participants whose best response is partial response (PR) or complete response (CR). | Day 22-29, every other month.

SECONDARY OUTCOMES:
Area under the plasma concentration curve (AUC) for ridaforolimus. | Part A, Cycle 0, Day 1 (pre-dose)
Area under the plasma concentration curve (AUC) for ridaforolimus. | Part A, Cycle 0, Day 5 (pre- and post-dose)
AUC for the ridaforolimus + MK-0752 doublet | Part A, Cycle 1, Day 1 (pre-dose)
AUC for the ridaforolimus + MK-0752 doublet | Part A, Cycle 1, Day 12 (pre- and post-dose)

REFERENCES:
- [Background] Piha-Paul SA, Munster PN, Hollebecque A, Argiles G, Dajani O, Cheng JD, Wang R, Swift A, Tosolini A, Gupta S. Results of a phase 1 trial combining ridaforolimus and MK-0752 in patients with advanced solid tumours. Eur J Cancer. 2015 Sep;51(14):1865-73. doi: 10.1016/j.ejca.2015.06.115. Epub 2015 Jul 18. PMID 26199039
- [Background] Gupta S, Argiles G, Munster PN, Hollebecque A, Dajani O, Cheng JD, Wang R, Swift A, Tosolini A, Piha-Paul SA. A Phase I Trial of Combined Ridaforolimus and MK-2206 in Patients with Advanced Malignancies. Clin Cancer Res. 2015 Dec 1;21(23):5235-44. doi: 10.1158/1078-0432.CCR-15-0180. Epub 2015 Jul 17. PMID 26187616